CLINICAL TRIAL: NCT06010225
Title: The Enhanced Recovery After Surgery (ERAS) Protocol Implementation in a National Tertiary-level Hospital: A Prospective Cohort Study
Brief Title: Effects of Implementing an ERAS Protocol
Status: Completed | Type: Observational
Sponsor: Ridho Ardhi Syaiful (Other)
Responsible Party: Sponsor-Investigator, Ridho Ardhi Syaiful, Medical Doctor, Digestive Surgery, Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Other Study IDs: DRCiptoMGH
Record Dates: First submitted 2023-07-18; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Enhanced Recovery After Surgery (ERAS) Protocol; Colorectal Surgery; Effectivity; Colorectal Neoplasms; Colorectal Cancer
Keywords: Enhanced Recovery After Surgery (ERAS) protocol; Outcome; colorectal surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group: Patients who met the inclusion criteria and consented were assigned to the ERAS group
- control group: Patients who met the inclusion criteria and did not consent were assigned to the ERAS group

SUMMARY:
Introduction: Successful colorectal surgery is determined based on postoperative mortality and morbidity rates, complication rates, and cost-effectiveness. One of the methods to obtain an excellent postoperative outcome is the Enhanced Recovery After Surgery (ERAS) protocol. This study aims to see the effects of implementing an ERAS protocol in colorectal surgery patients.

Methods: Eighty-four patients who underwent elective colorectal surgery at National Tertiary-level Hospital were included between January 2021 and July 2022. Patients were then placed into ERAS and control groups according to the criteria. The Patients in the ERAS group underwent a customized 18-component ERAS protocol and were assessed for adherence. Postoperatively, both groups were monitored for up to 30 days and assessed for complications and readmission. The investigators then analyzed the length of stay and total patient costs in both groups.

DETAILED DESCRIPTION:
The investigators aimed to determine whether applying the ERAS protocol to patients undergoing colorectal surgery could improve surgical outcomes (length of stay, complications, readmission, and total costs) in the National Tertiary Hospital clinical setting.

This prospective cohort study to analyze the implementation of ERAS protocol in colorectal patients and its effect on length of stay, readmission rate, complications, and costs in Dr. Cipto Mangunkusumo General Hospital, an Indonesian tertiary-level hospital, from January 2021 to July 2022. ERAS protocol used in this study was arranged based on the guidelines of the ERAS ® Society, with certain adjustments made to fit Indonesia's population characteristics. The sampling process was performed for all patients undergoing elective colorectal surgeries in The Central Surgery Room during the study period, who continued their medical care at Integrated Medical Ward Unit and fulfilled all inclusion and exclusion criteria. In this study, the investigators also used a multidisciplinary team approach that carried out various protocol points in all phases, according to their areas of expertise. This team comprised surgeons, anesthesiologists, physical medicine, internists, rehabilitation specialists, general physicians, dietitians, nurses, pharmacists, surgery admission staff, medical record staff, and hospital administration staff.

Study participants The investigators evaluated patients in two different groups: ERAS and non-ERAS. In both groups, the investigators included patients who underwent elective/non-emergency colorectal surgery above 18 years of age, with a maximum of two different comorbidities to minimize postoperative complications, a body mass index above 18.5 kg/m2, and an ASA below 2. In the ERAS group, patients were first evaluated for eligibility for the ERAS protocol and their willingness to follow a series of ERAS protocols at the outpatient clinic of the Cipto Mangunkusumo Hospital. The Patients registered in the ERAS group followed the protocol of the ERAS research team. For the control group, patients selected through examination in the outpatient clinic would undergo conventional/traditional surgery.

The sample size was calculated using an unpaired numerical, analytical research sample size formula, with an alpha of 5%, a beta of 10%, a combined standard deviation of four based on previous studies, and an assumed mean outcome difference of 3. To obtain a minimum sample size for each group of 37 subjects.

Outcomes The primary outcomes of this study were: (1) the length of hospitalization, (2) postoperative complications, (3) readmission rate, and (4) total medical costs. The length of hospitalization was calculated from the day of admission to the hospital ward until discharge. Postoperative complications were defined as infection on the surgical site or systemic infection, wound dehiscence, and other complications found after surgery. The readmission rate was calculated from discharge to one month after surgery. Total medical costs were calculated based on direct medical costs recorded in the hospital billing data. The currency was converted from Indonesian Rupiah (IDR) to US dollars (USD) based on the September 1, 2022, conversion rate of USD 1 = IDR 14,200.

In addition, the investigators assessed the adherence of patients in the ERAS group to the ERAS protocol. Each implemented protocol component was recorded, and the number of protocols that could be implemented for each patient was calculated. The adherence to the eighteen ERAS protocols was grouped into: <90%, 90-95%, 96-100% for readmission, complications, length of stay <7 days, and costs < USD 3,000 for patients in the ERAS group based on a previous study. The controlled price of USD 3,000 is determined based on hospital's average cost of the non-ERAS group.

ELIGIBILITY:
Inclusion Criteria:

* maximum of two different comorbidities
* body mass index above 18.5 kg/m2
* ASA below 2

Exclusion Criteria:

* More than 2 comorbidities
* Refused to take part in the research

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients undergoing surgery at Dr. Cipto Mangunkusumo General Hospital
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
length of hospitalization | day 1 until day 30
  The length of hospitalization was calculated from the day of admission to the hospital ward until the discharge
postoperative complications | day 1 until day 30
  Postoperative complications were defined as infection on the surgical site or systemic infection, wound dehiscence, and other complications found after surgery
readmission rate | day 1 until day 30
  The readmission rate was calculated from discharge to one month after surgery.
Total medical costs | day 1 until day 30
  Total medical costs were calculated based on direct medical costs recorded in the hospital billing data. The currency was converted from Indonesian Rupiah (IDR) to US dollars (USD) based on the September 1, 2022, conversion rate of USD 1 = IDR 14,200.

SECONDARY OUTCOMES:
adherence to the ERAS protocols | day 1 until day 30
  The adherence to the eighteen ERAS protocols was grouped into: <90%, 90-95%, 96-100% for readmission, complications, length of stay <7 days, and costs < USD 3,000 for patients in the ERAS group based on a previous study

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Andreoni B, Chiappa A, Bertani E, Bellomi M, Orecchia R, Zampino M, Fazio N, Venturino M, Orsi F, Sonzogni A, Pace U, Monfardini L. Surgical outcomes for colon and rectal cancer over a decade: results from a consecutive monocentric experience in 902 unselected patients. World J Surg Oncol. 2007 Jul 4;5:73. doi: 10.1186/1477-7819-5-73. PMID 17610720
- [Background] Tevis SE, Kennedy GD. Postoperative Complications: Looking Forward to a Safer Future. Clin Colon Rectal Surg. 2016 Sep;29(3):246-52. doi: 10.1055/s-0036-1584501. PMID 27582650
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Alves A, Panis Y, Mathieu P, Mantion G, Kwiatkowski F, Slim K; Association Francaise de Chirurgie. Postoperative mortality and morbidity in French patients undergoing colorectal surgery: results of a prospective multicenter study. Arch Surg. 2005 Mar;140(3):278-83, discussion 284. doi: 10.1001/archsurg.140.3.278. PMID 15781793
- [Background] Tan JKH, Ang JJ, Chan DKH. Enhanced recovery program versus conventional care after colorectal surgery in the geriatric population: a systematic review and meta-analysis. Surg Endosc. 2021 Jun;35(6):3166-3174. doi: 10.1007/s00464-020-07673-7. Epub 2020 May 28. PMID 32468264
- [Background] Miller TE, Thacker JK, White WD, Mantyh C, Migaly J, Jin J, Roche AM, Eisenstein EL, Edwards R, Anstrom KJ, Moon RE, Gan TJ; Enhanced Recovery Study Group. Reduced length of hospital stay in colorectal surgery after implementation of an enhanced recovery protocol. Anesth Analg. 2014 May;118(5):1052-61. doi: 10.1213/ANE.0000000000000206. PMID 24781574
- [Background] Li L, Jin J, Min S, Liu D, Liu L. Compliance with the enhanced recovery after surgery protocol and prognosis after colorectal cancer surgery: A prospective cohort study. Oncotarget. 2017 Jun 22;8(32):53531-53541. doi: 10.18632/oncotarget.18602. eCollection 2017 Aug 8. PMID 28881829